CLINICAL TRIAL: NCT01253746
Title: Genetics of Neural Tubes Defects
Brief Title: Genetics of Neural Tube Defects
Acronym: NTD
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: John P. Hussman Institute for Human Genomics (Other)
Collaborators: University of Miami (Other)
Responsible Party: Evadnie Rampersaud, University of Miami John P. Hussman Institute for Human Genomics
Other Study IDs: 1072
Record Dates: First submitted 2010-12-02; First posted 2010-12-03 (Estimated); Last update posted 2010-12-03 (Estimated); Status verified 2010-12

CONDITIONS: Neural Tube Defects
Keywords: NTD; open NTD; spina bifida; anencephaly; closed NTD; lipomeningocele; tethered cord.
MeSH Terms: conditions — Neural Tube Defects; Spinal Dysraphism; Anencephaly; Spinal Cord Injuries

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood sample
Oversight: Data Monitoring Committee: No

SUMMARY:
The Genetics of Neural Tube Defects Study at the University of Miami: The University of Miami John P. Hussman Institute for Human Genomics is looking for families to participate in research to identify the genetic and environmental factors that contribute to Neural Tube Defects (NTD). Our research goal is to better understand the genetic and environmental causes of both open NTD, like spina bifida and anencephaly, and closed NTD, like lipomeningocele and tethered cord. This will eventually lead to more accurate genetic counseling and risk assessment, improved treatments, and better prevention methods. Any individual with a diagnosis of NTD and his/her selected family members can participate, if willing. Participation is free. Travel is not required. Participation involves reading and signing a consent form, providing a blood sample, a family and medical history interview, and granting the research staff permission to review the medical records of the individual(s) with NTD. We maintain the highest standards of confidentiality for all families. If interested, please contact Maria Ciliberti, the study coordinator, at 1-877-686-6444 (toll free) or directly at 305-243-4360, or by email Mciliberti@med.miami.edu . Please visit our web site at www.hihg.org for more information.

ELIGIBILITY:
Inclusion Criteria: Any individual with a diagnosis of NTD and his/her selected family members can participate, if willing -

Exclusion Criteria: Pregnant children will not be enrolled

-

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Any individual with a diagnosis of NTD and his/her selected family members can participate, if willing
Sampling Method: Non-Probability Sample
Enrollment: 6000 (Estimated)
Dates: Start 2009-04

CONTACTS AND LOCATIONS:
Overall Officials: Evadnie Rampersaud, PhD, Principal Investigator — University of Miami John P. Hussman Institute for Human Genomics
Locations (1):
- University of Miami John P. Hussman Institute for Human Genomics, Miami, Florida, United States

REFERENCES:
- See also: Related Info — http://hihg.org